CLINICAL TRIAL: NCT03407898
Title: The Effect of Different Videolaryngoscopes on Intubation Success in Difficult Airway Patients
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Associated professor, Ankara University
Other Study IDs: 20-1006-16
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Mallampati Score, Difficult Intubation, Videolaryngoscope

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C-mac D blade used for intubation
  Interventions: Other: intubation time
- mcgrath X blade used for intubation
  Interventions: Other: intubation time

INTERVENTIONS:
Other: intubation time — intubation attempt number and intubation time
  Other Names: intubation attempt

SUMMARY:
Mallampati score > 3 generally indicate difficult airway and difficult intubation. Most anesthesiologist usually use this score system to predict difficult airway management. Different laryngoscopes may be useful in management of difficult airway. This study designed to compare different videolaryngoscopes in intubation success in patient of Mallampati score>3.

ELIGIBILITY:
Inclusion Criteria:

* mallampati score >3

Exclusion Criteria:

* patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who has mallampati score >3
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
intubation time | 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIMGUCLU, Study Chair — Ankara University
Locations (1):
- Cigdem Yildirimguclu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No